CLINICAL TRIAL: NCT05978349
Title: Vitro 3D Drug Sensitivity Detection of Micro Tumor (PTC) to Guide Postoperative Adjuvant Treatment Strategy and Prognosis Judgment of Colorectal Cancer--Prospective Clinical Study
Brief Title: PTC Drug Sensitivity Detection to Guide Postoperative Adjuvant of Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-PUMCH-B-005
Record Dates: First submitted 2023-07-27; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Colo-rectal Cancer
Keywords: colon cancer; rectal cancer; adjuvant therapy; PTC
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — In Vitro Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Select adjuvant chemotherapy scheme according to 3D drug sensitivity test results of micro tumor (PTC) in vitro
  Interventions: Drug: adjuvant therapy based on 3D drug sensitivity test results of micro tumor (PTC) in vitro
- control group (No Intervention): Formulate adjuvant chemotherapy strategy based on clinical experience

INTERVENTIONS:
Drug: adjuvant therapy based on 3D drug sensitivity test results of micro tumor (PTC) in vitro — Choose chemotherapeutic drugs（5-fluorouracil + formyltetrahydrofolate/Oxaliplatin + 5-fluorouracil + formyltetrahydrofolate/Irinotecan + 5-fluorouracil + formyltetrahydrofolate/Cetuximab + 5-fluorouracil + formyltetrahydrofolate） based on PTC drug sensitivity results.
  Other Names: PTC drug sensitivity results
  Arms: experimental group

SUMMARY:
The research objectives is to compare vitro 3D drug sensitivity test results of micro tumor (PTC) with the clinical outcomes of patients, evaluate the consistency between the test results of the technology platform and the clinical prognosis, and explore the decision-making value and guiding significance of this technology in assisting the precise treatment of colorectal cancer. The completion of this study will provide real-world data support for the clinical application of micro tumor (PTC) in vitro 3D drug sensitivity detection technology, and provide more valuable reference basis for realizing the individualization and accuracy of colorectal cancer treatment and improving the clinical benefit rate.

DETAILED DESCRIPTION:
The study is a multi agency prospective cohort study in China. The subjects were patients aged 18 ~ 75 years with colorectal cancer diagnosed by histopathology or cytology. They must be colorectal cancer patients who have at least one assessable tumor focus, need adjuvant therapy after radical surgery, and have not received neoadjuvant therapy， ECoG physical condition score ≤ 2 points. And they must be voluntarily participate in and sign informed consent.

The patients were randomly divided into PTC drug sensitivity test group and control group. The PTC drug sensitivity test group selected the adjuvant chemotherapy scheme according to the 3D drug sensitivity test results of micro tumor (PTC) in vitro. The control group made adjuvant chemotherapy strategy according to clinical experience.

The primary endpoint was the non inferiority test, and the 3-year disease-free survival rate was T-C >- Δ

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 75 years old, regardless of gender
2. Patients with colorectal cancer diagnosed by histopathology or cytology
3. Colorectal cancer patients who need adjuvant therapy after radical surgery and have not received neoadjuvant therapy
4. Having at least one assessable tumor focus
5. ECoG physical condition score ≤ 2 points
6. Voluntarily participate and sign informed consent

Exclusion Criteria:

1. Patients diagnosed with metastasis
2. Patients who cannot obtain tumor samples
3. Pregnant and lactating women
4. Patients with poor compliance
5. Patients with severe cardiovascular and cerebrovascular complications who cannot receive adjuvant treatment
6. Patients with other malignant tumors
7. Suffering from serious mental and nervous system diseases
8. The researchers believe that patients should not be selected for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Follow-up and record DFS of patients | 3 years after enrollment
  We follow-up the patients by outpatient/telephone/online message to find out their survival situation and record their Disease-free-survival time

SECONDARY OUTCOMES:
Follow-up and record TTP of patients | 3 years after enrollment
  We follow-up the patients by outpatient/telephone/online message to find out their tumor situation and record their Time To Progress
Consistency between drug sensitivity results and clinical outcomes | 3 years after enrollment
  Record the patient's PTC drug sensitivity results and the actual medication therapy, and record the patient's survival status through telephone follow-up, online follow-up and offline diagnosis to compare whether there is correlation between them.
Follow-up and record ORR of patients | 3 years after enrollment
  We follow-up the patients by outpatient/telephone/online message to find out their tumor situation and record their Objective Response Rate
Follow-up and record PFS of patients | 3 years after enrollment
  We follow-up the patients by outpatient/telephone/online message to find out their tumor situation and record their Progress Free Survival time
Follow-up and record OS of patients | 3 years after enrollment
  We follow-up the patients by outpatient/telephone/online message to find out their tumor and survival situation and record their Overall Survival time

CONTACTS AND LOCATIONS:
Overall Officials: Guo Lin, Professor, Study Chair — PUMCH
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, China/Beijing, China

IPD SHARING:
Plan to Share IPD: No